CLINICAL TRIAL: NCT05911828
Title: Phase Ib, Single-center, Randomized, Study to Determine Safety, Tolerability, and Pharmacokinetics of Different Orally Administered Regimens of the Combination ZY19489-Ferroquine in Adult Asymptomatic Plasmodium Falciparum Carriers
Brief Title: A Study to Determine Safety, Tolerability, and Pharmacokinetics of Different Orally Administered Regimens of the Combination ZY19489-Ferroquine in Adult Asymptomatic Plasmodium Falciparum Carriers
Acronym: ZYFER-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZY-19489.23.001
Record Dates: First submitted 2023-06-04; First posted 2023-06-22 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Uncomplicated Malaria; Asymptomatic Condition; Falciparum Malaria
MeSH Terms: conditions — Asymptomatic Diseases; Malaria, Falciparum | interventions — ZY-19489; ferroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZY19489 + Ferroquine (FQ) (Active Comparator): A single daily dose 600 mg ZY19489 + 600 mg FQ, or 900 mg ZY19489 + 900 mg FQ are selected as the doses to be evaluated in Cohort 1 and 2, respectively. A daily dose of 600 mg ZY19489 + 600 mg FQ will be administered daily for 2 days in Cohort 3.
  ZY19489-FQ combination or placebo orally after a fasting period of at least 10 h.
  Interventions: Drug: ZY19489 + Ferroquine (FQ)
- Placebo (Placebo Comparator): ZY19489-FQ combination or placebo orally after a fasting period of at least 10 h.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZY19489 + Ferroquine (FQ) — ZY19489-FQ combination or placebo orally after a fasting period of at least 10 h.
  Arms: ZY19489 + Ferroquine (FQ)
Drug: Placebo — ZY19489-FQ combination or placebo orally after a fasting period of at least 10 h.
  Arms: Placebo

SUMMARY:
Malaria is caused by protozoan parasites of the genus Plasmodium and it is the most important parasitic disease in terms of mortality and morbidity. Estimates of 247 million malaria cases and 619.000 deaths worldwide were reported by WHO for the year 2021 (1). Plasmodium falciparum can lead to severe malaria and accounts for 90% of malaria deaths that mainly occur in children below the age of 5 years in Sub-Saharan Africa.

A simplified treatment regimen, ideally a single-day cure (or at most 2-day dosing regimen), of uncomplicated malaria due to P. falciparum would be the magic in the antimalarial armamentarium. Improving treatment adherence is one of the key factors in reducing mortality and morbidity and also the transmission of malaria, and such a regimen would substantially increase adherence. To find a new non-artemisinin combination therapy with a shorter regimen, ideally, a single-dose cure, with low resistance potential would be the aim. The two compounds tested here are ZY19489, a triaminopyrimidine, and ferroquine (FQ), a next-generation 4-aminoquinoline. Both compounds show unique features in terms of long half-life, and activity against current drug-resistant strains.

Therefore, the main goal of this clinical trial is to assess the safety of the ZY19489-FQ combination given as a 1- or 2-day dose regimen.

DETAILED DESCRIPTION:
Total of 36 participants (3 cohorts with up to 12 participants each).The participant will receive the intervention orally once daily for one or two days, following a fasting period of at least 10 hours.Total duration of trial participation for each participant: Approximately 10 weeks (screening visits + 64 days of follow-up).

ELIGIBILITY:
Inclusion Criteria:

- 1. Male and female (non-pregnant, non-lactating) subjects aged between 18 and 55 years old 2. Participant's body weight ≥ 45 kg 3. Evidence of asymptomatic infection with Plasmodium falciparum mono-infection on microscopy with parasite density between 20/µL and 5000/µL.

4. Participants should agree to not donate blood from enrolment in the study until end of the follow-up period 5. Ability to swallow oral medication 6. Evidence of written informed consent personally signed and dated by the participant.

Signed informed consent obtained prior to participation in the study. In case of participant unable to read and write or otherwise incapable of signing an informed consent, an impartial witnessed consent shall be obtained. Participants who are willing to and are able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* 1. Mixed Plasmodium infection as judged by microscopy. 2. Presence of clinically significant infectious disease or fever (e.g. Body temperature ≥38°C or 100.4°F) within the 14 days prior to enrollment.

  3. History of alcohol or drug abuse or positive urine alcohol test or urine drug test.

  4. Consumption of beverages or food containing xanthine bases including chocolate, coffee etc. from 48 hours prior to enrollment.

  5. Known allergy to the study drugs and to the rescue medications (artemisinin derivatives, lumefantrine) as well as their excipients.

  6. History of having received any antimalarial treatment (alone or in combination) during the following periods before screening:
  1. Piperaquine, mefloquine, naphthoquine or sulfadoxine-pyrimethamine within 6 weeks prior to screening.
  2. Amodiaquine, chloroquine within 4 weeks prior to screening.
  3. Any artemisinin derivative (artesunate, artemether or dihydroartemisinin), quinine, lumefantrine or any other anti-malarial treatment or antibiotic with antimalarial activity (including cotrimoxazole, tetracyclines, quinolones and fluoroquinolones and azithromycin) within 14 days prior to screening.

     7. Laboratory parameters outside normal range or with clinically relevant abnormalities as per investigator's judgment.

     8. Electrolyte levels outside normal range 9. Hematology, clinical chemistry or urinalysis results at screening that were outside of clinically acceptable laboratory ranges and were considered clinically significant by the Investigator.

     10. GFR<60 ml/min. 11. Previous participation in any malaria vaccine study or received malaria vaccine in any other circumstance within 3 months of screening.

     12. Participation in other clinical studies within 90 days before screening. 13. Pregnant or nursing (lactating) women. 14. Sexually active participants not willing to take effective contraception measures from enrolment until the last study visit: For female participants, combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner.

     15. All male participants not willing to use either true abstinence, barrier method or with their sexual partner, the use of effective means of contraception from enrolment and until the last study visit.

     16. Participant who the investigator considers at particular risk of receiving an anti-malarial or of participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
incidence, severity and relationship to ZY19489-FQ of treatment emergent adverse events | Day 0 to Day 64
  To evaluate the safety and tolerability of ZY19489-FQ combination in African adult asymptomatic carriers of Plasmodium falciparum mono-infections.

SECONDARY OUTCOMES:
Area under the curve from the time of dosing to the last measurable concentration (AUC0-t). | Day 0 to Day 64
  Estimation of PK parameters of ZY19489, its major metabolite and FQ and its major metabolite using noncompartmental method.To characterize the PK of ZY19489-FQ combination in African asymptomatic adult carriers of Plasmodium falciparum mono-infections
Area under the curve from the time of dosing to the infinity (AUC0-∞) | Day 0 to Day 64
  Estimation of PK parameters of ZY19489, its major metabolite and FQ and its major metabolite using noncompartmental method.To characterize the PK of ZY19489-FQ combination in African asymptomatic adult carriers of Plasmodium falciparum mono-infections
Maximum plasma concentration (Cmax) | Day 0 to Day 64
  Estimation of PK parameters of ZY19489, its major metabolite and FQ and its major metabolite using noncompartmental method.To characterize the PK of ZY19489-FQ combination in African asymptomatic adult carriers of Plasmodium falciparum mono-infections
Time to reach maximum plasma concentration (Tmax) | Day 0 to Day 64
  Estimation of PK parameters of ZY19489, its major metabolite and FQ and its major metabolite using noncompartmental method.To characterize the PK of ZY19489-FQ combination in African asymptomatic adult carriers of Plasmodium falciparum mono-infections
Terminal half life (t1/2) | Day 0 to Day 64
  Estimation of PK parameters of ZY19489, its major metabolite and FQ and its major metabolite using noncompartmental method.To characterize the PK of ZY19489-FQ combination in African asymptomatic adult carriers of Plasmodium falciparum mono-infections
Clearance (CL/F) | Day 0 to Day 64
  Estimation of PK parameters of ZY19489, its major metabolite and FQ and its major metabolite using noncompartmental method.To characterize the PK of ZY19489-FQ combination in African asymptomatic adult carriers of Plasmodium falciparum mono-infections
Volume of distribution (Vd/F) | Day 0 to Day 64
  Estimation of PK parameters of ZY19489, its major metabolite and FQ and its major metabolite using noncompartmental method.To characterize the PK of ZY19489-FQ combination in African asymptomatic adult carriers of Plasmodium falciparum mono-infections
Elimination rate constant (λ) | Day 0 to Day 64
  Estimation of PK parameters of ZY19489, its major metabolite and FQ and its major metabolite using noncompartmental method.To characterize the PK of ZY19489-FQ combination in African asymptomatic adult carriers of Plasmodium falciparum mono-infections

OTHER OUTCOMES:
Parasite reduction ratio between baseline and 48h post-treatment (PRR48) and corresponding parasite clearance half-life (PCT½). | Day 0 to Day 64
  To describe the parasite clearance capacity of ZY19489-FQ combination in African asymptomatic adult carriers of Plasmodium falciparum mono-infections

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Deven Parmar, MD,FCP, Study Director — Zydus Therapeutics Inc.
Locations (1):
- Centre de Recherches Médicales de Lambaréné, Lambaréné, Gabon

IPD SHARING:
Plan to Share IPD: No